CLINICAL TRIAL: NCT05053451
Title: Transcranial Direct Current Stimulation (tDCS) Studies of Auditory Hallucinations, Negative Symptoms and Cognition in Schizophrenia
Brief Title: Brain Stimulation, Clinical Symptoms and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1607658
Record Dates: First submitted 2021-09-02; First posted 2021-09-22 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; EEG; tDCS; dorsolateral prefrontal cortex; temporoparietal junction; cognitive control; auditory hallucinations; transcranial direct current stimulation
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- dlPFC/TPJ Stimulation + Rest (Experimental): 20 minutes of 2 mA direct current stimulation during rest.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In tDCS, saline-soaked electrodes are temporarily affixed to the scalp and connected to a battery-powered current generator. A weak (2 mA) constant current is then briefly applied (20 minutes) to stimulate the targeted brain area (e.g. the DLPFC, TPJ, Occipital Cortex) depending on the phase of the study.

SUMMARY:
The purpose of this study is to test the impact of non-invasive brain stimulation, transcranial direct current stimulation (tDCS), on auditory hallucinations, negative symptoms and cognition in schizophrenia. Clinical measures will be used to assess clinical symptoms and cognitive performance to test the hypothesis that a course of tDCS can reduce auditory hallucinations and negative symptoms in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to sufficiently speak and understand English so as to be able to understand and complete cognitive tasks.
* All subjects must have the ability to give valid informed consent.
* No children under the age of 18 will be recruited.
* Diagnosis of schizophrenia, schizophreniform, or schizoaffective disorder
* Stable outpatient or partial hospital status
* Normal IQ (>70; IQ will be measured by administering the Wechsler Abbreviated Scale of Intelligence (WASI) test)

Exclusion Criteria:

* Pacemakers
* Implanted electrical (brain and spinal) stimulators
* Implanted defibrillator
* Metallic implants
* Skin damage or skin conditions such as eczema at the sites where electrodes will be placed
* Hair styles hindering the placement of electrodes
* Cranial pathologies
* Head trauma
* Epilepsy
* Mental retardation
* Any known history of neurological disorders (including epilepsy, amyotrophic lateral sclerosis (ALS), multiple sclerosis (MS), stroke, cerebral palsy, any DSM-5 axis I psychiatric disorder (for healthy control subjects), autism)
* Uncorrected vision problems that would hinder cognitive testing (this also pertains to subjects with color blindness in tasks where discriminating colored objects/items is necessary for successful performance)
* Pregnancy
* Substance dependence in the past six months
* Substance abuse in the past month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Change in Symptom Severity of Auditory Hallucinations | Assessment begins with the initial baseline interview and concludes after a 2-week follow-up assessment using the same clinical measures.
  Participants will undergo diagnostic (clinical) interviews to rate their symptom severity using measures including, but not limited to, the Brief Psychiatric Rating Scale (rated 1-7, with a high rating indicating more severe symptoms), the Scale of the Assessment of Positive Symptoms (rated 0-5, with a high rating indicating more severe symptoms), and the Scale for the Assessment or Negative Symptoms (rated 0-5, with a high rating indicating more severe symptoms).
Change in Symptom Severity of Negative Symptoms | Assessment begins with the initial baseline interview and concludes after a 2-week follow-up assessment using the same clinical measures.
  Participants will undergo diagnostic (clinical) interviews to rate their symptom severity using measures including, but not limited to, the Brief Psychiatric Rating Scale (rated 1-7, with a high rating indicating more severe symptoms), the Scale of the Assessment of Positive Symptoms (rated 0-5, with a high rating indicating more severe symptoms), and the Scale for the Assessment or Negative Symptoms (rated 0-5, with a high rating indicating more severe symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Imaging Research Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Select data from this study may be submitted to the National Institute of Mental Health Data Archive (NDA). NDA is a data repository run by the National Institute of Mental Health (NIMH) that allows researchers studying mental illness to collect and share de-identified information with each other. The data repository is accessible only to qualified investigators. All subject data will be de-identified (subject names will not be used) and each subject will have a separate identifier called a Global Unique Identifier (GUID) to remove any possibility that "the identities of the subjects cannot be readily ascertained or otherwise associated with the data by the repository staff or secondary data users." (45 CFR, 46.102).